CLINICAL TRIAL: NCT04254250
Title: Observational Cohort Study Of The Efficacy Of Preoperative Estimation Of Disc Herniation Recurrence In Patients With Lumbar Disc Herniation
Brief Title: Preoperative Estimation Of Disc Herniation Recurrence In Patients With Lumbar Disc Herniation
Status: Active, not recruiting | Type: Observational
Sponsor: Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan (Other Government)
Responsible Party: Sponsor
Other Study IDs: NS02-03
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Intervertebral Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High risk recurrence group: Due to preoperative risk estimation each patient will be assigned to one of two groups - with high risk and low risk.
  Interventions: Diagnostic Test: Preoperative risk estimation of disc herniation recurrence
- Low risk recurrence group: Due to preoperative risk estimation each patient will be assigned to one of two groups - with high risk and low risk.
  Interventions: Diagnostic Test: Preoperative risk estimation of disc herniation recurrence

INTERVENTIONS:
Diagnostic Test: Preoperative risk estimation of disc herniation recurrence — Risk estimation of disc herniation recurrence will be evaluated preoperatively, depend on the risk significance each patient will be assigned to one of two groups - with high risk and low risk. Then each patient will undergo conventional one-level microdiscectomy.

SUMMARY:
This study will be conducted at Research Institute of Traumatology and Orthopedics (NRITO) n.a. Ya.L.Tsivyan, Novosibirsk, Russia.

The current study is prospective observational study to evaluate the efficacy of preoperative estimation of disc herniation recurrence among patients with lumbar disc herniation using predictive mathematical model at terms 3 years postoperatively .

It is expected to enroll 350 patients aged 18-70 with lumbar disc herniation. Risk estimation of disc herniation recurrence will be evaluated preoperatively, then patient will undergo conventional microdiscectomy. Postoperative eximanation will include Visits every 6-months during 3 years to evaluate clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Age 18 to 60 years;

Single level lumbar disc herniation with neural compression confirmed on MRI at one level of L4-L5 or L5-S1;

1. Radicular leg pain with or without back pain;
2. Symptoms persisting for at least four weeks prior to surgery;
3. Given written Informed Consent;
4. Able and agree to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements;
5. Visual Analogue Scale score at least 40/100 at baseline.

Exclusion Criteria:

1. More than one symptomatic level requiring multilevel surgical decompression
2. Stenosis any etiology at the same level;
3. Spondylolisthesis any etiology at the same level;
4. Prior lumbar spinal surgery at any level;
5. Other non-degenerative spinal conditions (e.g. infectious, traumatic, metabolic, inflammatory, neoplastic, structural or other pathology) that may have an impact on subject safety, wellbeing or the intent and conduct of the study
6. Concurrent participation in another clinical study that may confound study results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with radicular leg pain with or without back pain secondary to single level disc herniation with neural compression confirmed on MRI and symptoms persisting for at least four weeks prior to surgery
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Reherniation rate | at 3 years follow-up term postoperatively
  Rate of lumbar disc reherniation, symptomatic presence of disc herniation confirmed by MRI at the previously operated level and side

SECONDARY OUTCOMES:
Improvement of Oswestry Disability Index (ODI) | 6, 12, 18, 24, 30, 36 months follow up
  To observe the improvement of ODI as compared to baseline through follow-up terms Oswestry Disability Index - patient-reported physical and household activity. Minimum - 0 % (the best result, the patient has no limitations in physical activity). Maximum - 100% (the worst result, patient is not physically active at all).
Improvement of Visual analog scale (VAS) leg pain intensity | 6, 12, 18, 24, 30, 36 months follow up
  To observe the improvement of VAS leg pain as compared to baseline through follow-up terms.
Change from baseline in EQ-5D (EuroQl - 5 dimensional) | 6, 12, 18, 24, 30, 36 months follow up
  To observe change in EQ-5Dl as compared to baseline
HTI Item (from SF-36) | 6, 12, 18, 24, 30, 36 months follow up
  To observe the HTI Item (from SF-36) as compared to baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Priorov National Medical Research Center of Traumatology and Orthopedics, Moscow
  - Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan, Novosibirsk